CLINICAL TRIAL: NCT06200207
Title: Effects of Ziltivekimab Versus Placebo on Heart Failure Symptoms and Physical Function in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction and Systemic Inflammation
Brief Title: A Research Study Looking Into How Ziltivekimab Works Compared to Placebo in Participants With Heart Failure and Inflammation
Acronym: ATHENA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6018-4914; U1111-1293-7516 (Other: World Health Organisation (WHO)); 2023-506988-34 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Systemic Inflammation
MeSH Terms: conditions — Heart Failure | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ziltivekimab (Active Comparator): Participants will receive ziltivekimab administered subcutaneously (s.c.) once-monthly and added to standard of care for 12 months.
  Interventions: Drug: Ziltivekimab
- Placebo (Placebo Comparator): Participants will receive placebo matched to ziltivekimab administered s.c. once-monthly and added to standard of care for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Zilitivekimab will be administered subcutaneously once-monthly.
  Arms: Ziltivekimab
Drug: Placebo — Placebo matched to ziltivekimab will be administered subcutaneously once-monthly.
  Arms: Placebo

SUMMARY:
The study is being done to see if ziltivekimab can be used to treat participants living with heart failure and inflammation. Participants will either get ziltivekimab (active medicine) or placebo (inactive substance that looks like the study medicine but does not contain any medicine). The treatment participants get is decided by chance. Participant's chance of getting ziltivekimab or placebo is the same. Ziltivekimab is not yet approved in any country or region in the world. It is a new medicine that doctors cannot prescribe. The study is expected to last for up to 1 year and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Serum high-sensitivity C-reactive protein (hs-CRP) greater than or equal to 2 milligrams per liter (mg/L) at screening (visit 1)
* Disease specific - cardiovascular:
* N-terminal-pro-brain natriuretic peptide (NT-proBNP) greater than or equal to 225 picograms per milliliter (pg/mL) (375 pg/mL for participants with atrial fibrillation/flutter) at screening
* Diagnosis of heart failure (New York heart association (NYHA) Class II-III)
* Left ventricular ejection fraction (LVEF) greater than 40 percent documented by echocardiography within 12 months prior to or at screening (visit 1). The LVEF must be documented in medical records and the most recent measurement must be used to determine eligibility with no interim event signalling potential deterioration in ejection fraction (example myocardial infarction (MI) or heart failure (HF) hospitalisation)
* Structural heart disease and/or functional heart disease documented by echocardiography within 12 months prior to or at screening (visit 1) showing at least one of the following:

  1. Left atrial (LA) volume index greater than 34 milliliter per square meter (mL/m^2)
  2. LA diameter greater than or equal to 3.8 centimeter (cm)
  3. LA length greater than or equal to 5.0 cm
  4. LA area greater than or equal to 20 square centimeter (cm^2)
  5. LA volume greater than or equal to 55 milliliter (mL)
  6. Intraventricular septal thickness greater than or equal to 1.1 cm
  7. Posterior wall thickness greater than or equal to 1.1 cm
  8. LV mass index greater than or equal to 115 gram per square meter (g/m^2) in men or greater than or equal to 95 g/m^2 in women

  h) E/e' (mean septal and lateral) greater than or equal to 10 i) e' (mean septal and lateral) less than 9 centimeter per second (cm/s)
* No heart failure hospitalisations or urgent heart failure visits between screening and randomisation
* Able to perform the 6-minute walk test (6MWT) at screening with a minimum distance of 100 metres
* Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score lesser than 80 at screening

Exclusion Criteria:

* Medical conditions - cardiovascular:
* Myocardial infarction, stroke, unstable angina pectoris, transient ischaemic attack, or heart failure hospitalisation within 30 days prior to screening (visit 1)
* Systolic blood pressure greater than or equal to 180 millimeters of mercury (mmHg) at screening (visit 1). If the systolic blood pressure is 160-179 mmHg, the patient should be receiving greater than or equal to 3 antihypertensive drugs
* Heart rate above 110 or below 40 beats per minute as evaluated on the Electrocardiogram (ECG) performed at screening (visit 1)
* Planned coronary, carotid or peripheral artery revascularisation known during the screening period (visit 1)
* Planned cardiac device or atrial flutter/atrial fibrillation ablation procedure known during the screening period (visit 1)
* Major cardiac surgical, non-cardiac surgical, or major endoscopic procedure (thoracoscopic or laparoscopic) within the past 60 days prior to randomisation (visit 2) or any major surgical procedure planned at the time of randomisation (visit 2)
* Heart failure due to infiltrative cardiomyopathy (e.g., sarcoid, amyloid), arrhythmogenic right ventricular cardiomyopathy, Takutsubo cardiomyopathy, genetic hypertrophic cardiomyopathy or obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac tamponade, uncorrected more than moderate primary valve disease
* Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease including chronic obstructive pulmonary disease (COPD)
* Any other condition judged by the investigator that could account for heart failure symptoms and signs (e.g., anaemia, hypothyroidism)
* Medical conditions - infections/immunosuppression:
* Clinical evidence of, or suspicion of, active infection at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score (KCCQ-CSS) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as score (score on scale; range; 0-100). The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.

SECONDARY OUTCOMES:
Participant achieving threshold for clinically meaningful within-participant change in KCCQ CSS (yes/no) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as count of participants. The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Participant achieving threshold for clinically meaningful within-participant change in 6-minute walk distance (6MWD) (yes/no) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as count of participants.
Participants improving 5 points or more in KCCQ-CSS (yes/no) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as count of participants. The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Participants improving 10 points or more in KCCQ-CSS (yes/no) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as count of participants. The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Change in subscales of KCCQ (total symptom score, physical limitations score, social limitations score, and health-related quality of life) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as score (score on scale; range 0-100). The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Change in six-minute walk distance (6MWD) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured in meters.
Change in high-sensitivity C-reactive protein (hs-CRP) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as ratio to baseline.
Participants experiencing improvement in New York heart association (NYHA) Class (yes/no) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as count of participants. The New York Heart Association (NYHA) classification provides a simple way of classifying the extent of heart failure (HF). It classifies patients in one of four categories based on their limitations during physical activity - Class I: Participant with cardiac disease but without resulting limitations of physical activity, Class II: Participants with cardiac disease resulting in slight limitation of physical activity, Class III: Participants with cardiac disease resulting in marked limitation of physical activity, Class IV: Participants with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Change in N-terminal-pro-brain natriuretic peptide (NT-proBNP) | From randomisation (month 0) to end-of-treatment (month 12)
  Measured as ratio to baseline.
Change in eGFR (CKD-EPI) | From randomisation (month 0) to end-of-treatment (month 12)
  eGFR (CKD-EPI) is estimated glomerular filtration rate chronic kidney disease - epidemiology collaboration. Measured in milliliter per minute per 1.73 square meter (ml/min/1.73^2).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (211):
- United States (37):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Eastern Shore Rsrch Inst, LLC, Fairhope, Alabama
  - Cardiology & Medicine Clinic, Little Rock, Arkansas
  - Valley Clinical Trials, Inc., Northridge, California
  - UCI Health, Orange, California
  - South California Heart Spc, Pasadena, California
  - Clearwater Cardiovascular Consultants, Largo, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - St Johns Ctr Clin Rsch-St. Aug, Saint Augustine, Florida
  - GA Arrhythmia Cons & Rsch Inst, Macon, Georgia
  - Velocity Clin Rsrch - Savannah, Savannah, Georgia
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - UofL Health Care Outpatient, Louisville, Kentucky
  - Maryland Cardiovascular Specialists - Baltimore, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Cardio and Vascular Assoc-CAVA, Bloomfield Hills, Michigan
  - Millennium Cardiology, Farmington Hills, Michigan
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Long Island Cardiovascular Consultants PC, Lake Success, New York
  - Mount Sinai Hosp at NYC, New York, New York
  - Northwell Health Phys Cardio, Riverhead, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - AMS Cardiology, Horsham, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - PharmaTex Research, Amarillo, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - David Turbay, MD, PLLC, El Paso, Texas
  - Private Practice Leadership LLC., Katy, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - Clinical Advancement Ctr, PLLC, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Northwest Heart Center, Tomball, Texas
  - Sentara Health Research Center, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (10):
  - Cardiología Palermo, City of Buenos Aires, Buenos Aires
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Buenos Aires
  - CIPREC Pueyrredon, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, CABA
  - Sanatorio Esperanza, Esperanza, Santa Fe
  - Consultorio Integral de Atención al Diabético, Morón
  - Centro Cardiovascular Salta, Salta
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán.
- Australia (9):
  - Canberra Hospital, Garran, Australian Capital Territory
  - John Hunter Hospital - Cardiovascular Department, New Lambton Heights, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Illawarra Heart Health Centre, Wollongong, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Ballarat Base Hospital, Ballarat, Victoria
  - The Cardiologists Pty Ltd, Epping, Victoria
  - Advara HeartCare, Mulgrave, Victoria
  - Fiona Stanley Hospital Cardiology, Murdoch, Western Australia
- Bulgaria (9):
  - MHAT "Puls" AD Cardiology Department, Blagoevgrad
  - MHAT Haskovo AD, Haskovo
  - MHAT Heart and Brain, Pleven
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Cardiology, Plovdiv
  - "Medical Center Hera" EOOD - Sofia, Sofia
  - Medical center ISUL - Tsaritsa Yoanna EOOD, Sofia
  - UMHATEM N.I. Pirogov EAD, Sofia
  - UMHAT Sveta Anna Sofia AD, Clinic of Cardiology, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
- Canada (10):
  - University of Calgary_Calgary, Calgary, Alberta
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Saul Vizel Pro. Med. Corp, Cambridge, Ontario
  - Corcare Cardiovascular Research, Scarborough Village, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - CPS Research, Waterloo, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - CHU de Quebec-Uni Laval-Hotel, Québec
- Czechia (8):
  - Innera s.r.o., Benešov
  - Kardiologicka ambulance Brno s.r.o., Brno
  - Vojenská nemocnice Brno p.o., Brno
  - Ordinace pro choroby srdce, Chomutov
  - MEDICON a.s., Prague
  - Svitavska nemocnice Kardiologie, Svitavy
  - Kardiologie Trutnov Ferkl, Trutnov
  - Nemocnice AGEL Třinec-Podlesí a.s., Třinec
- France (7):
  - Centre Hospitalier Regional Universitaire de Tours-Hopital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen-Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Intercommunal Toulon La Seine-Sur-Mer - Hopital Sainte Musse, Toulon
  - Polyclinique Vauban, Valenciennes
  - Chru de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (10):
  - Kardiologisch-Angiologische Praxis Herzzentrum Bremen, Bremen
  - Uniklinik TU Dresden - Herzzentrum Dresden GmbH, Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - Kath. Hospitalvereinigung Thüringen gGmbH - KKH St. Johann Nepomuk - Innere Med. II, Erfurt
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau
  - MVZ im Altstadt-Carree Fulda GmbH - Zentrum für klinische Studien, Fulda
  - Universität des Saarlandes - Innere Med. III, Homburg
  - Kardiopraxis Schirmer, Kaiserslautern
  - Gesundheitscentrum Mainz (Regner / Schmitt), Mainz
- Greece (18):
  - Alexandra General Hospital, Therapeutic Clinic, Athens, Attica
  - Evangelismos Hospital, Athens
  - Naval Hospital of Athens - Clinic of Cardiology, Athens
  - "Laiko" General Hospital of Athens, Athens
  - 'G. Gennimatas' General Hospital of Athens - Cardiology Department, Athens
  - 'G. Gennimatas' General Hospital of Athens, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - Metropolitan General Hospital Healthcare Facilities Operation And Management Single Member S.A. - Cardiology Clinic, Athens
  - Naval Hospital of Athens, Athens
  - U.G.H of Athens "Attikon", Chaidari, Athens
  - General Hospital of Kalamata - Cardiology Department, Chalcis
  - General Hospital of Chios "Skilitsio" - Cardiology Clinic, Chios
  - Univ Gen Hospital Larisa, Cardiology Medicine Clinic, Larissa
  - Sismanogleio General Hospital - Cardiology Department, Marousi
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
  - Gen Hospital of Thessaloniki G.Papanikolaou,Cardiology Dpt, Thessaloniki
- India (29):
  - Siddhartha Medical College & Government General Hospital, Vijaywada, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Rhythm Heart Institute, Vadodara, Gujarat
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - KLES Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - St John's Medical College Hospital, Bengaluru, Karnataka
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bengaluru, Karnataka
  - Manipal Hospital, Mysuru, Mysuru, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Udupi, Karnataka
  - Sengupta Hospital and Research Institute, Nagpur, Maharashtra
  - All India Institute of Medical Sciences (AIIMS), Nagpur, Nagpur, Maharashtra
  - Chopda Medicare and Research Centre Pvt. Ltd., Nashik, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - Villoo Poonawalla Memorial Hospital, Pune, Maharashtra
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Vardhaman Mahavir Medical College & Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Bhubaneswar, Odisha
  - S.P. Medical College & Associated Group of Hospitals, Bikaner, Rajasthan
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry, Tamil Nadu
  - Guru Nanak CARE Hospitals, Hyderabad, Telangana
  - Malla Reddy Narayana Multispeciality Hospital, Hyderabad, Telangana
  - Ganesh Shankar Vidyarthe Memorial (GSVM) Medical College, Kanpur, Uttar Pradesh
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Jawaharlal Nehru Medical College and Hospital, Aligarh, Utter Pradesh
  - B M Birla Heart Research Centre, Kolkata, West Bengal
- Malaysia (8):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak
  - Hospital Serdang, Kajang, Selangor
- Poland (23):
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Kardio Life - Tomasz Borkowski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Kardio Life, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Cardiomedicum Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Linden sp. z o.o. sp. k., Krakow, Lesser Poland Voivodeship
  - Formed 2 Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Pratia S.A., Jelenia Góra, Lower Silesian Voivodeship
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej W Pulawach, Puławy, Lublin Voivodeship
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - Szpitale Pomorskie Sp. z o.o., Gdynia, Pomeranian Voivodeship
  - American Heart of Poland S.A., Bielsko-Biala
  - 10 Wojskowy Szpital Kliniczny z Poliklinika - Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Bydgoszczy, Bydgoszcz
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Trialmed Sp. z o. o., Piotrkow Trybunalski
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan
  - American Heart of Poland S.A., Tychy
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Lodz, Łódź Voivodeship
- Portugal (5):
  - CHTâmega e Sousa - Hospital Padre Américo, Guilhufe - Penafiel
  - CHLO, EPE - Hospital São Francisco Xavier, Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar de Setubal, Setúbal
- Spain (9):
  - Hospital Vithas Sevilla, Castilleja de la Cuesta, Andalusia
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hosp. Virgen del Camino_Sanlúcar_Medicina Interna, Sanlúcar de Barrameda
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Fundación para la Investigación del Hospital Clínico de Valencia (INCLIVA), Valencia
- Turkey (Türkiye) (14):
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Kardiyoloji, Eskişehir, Odunpazari
  - T.C. Saglık Bakanlıgı Adana Sehir Egitim ve Arastirma Hastan, Adana
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Adana
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Afyonkarahisar Sağlık Bilimleri Üniversitesi Sağlık Uygulama Ve Araştırma Merkezi- Kardiyoloji, Afyonkarahisar
  - Ankara Bilkent Şehir Hastanesi-Kardiyoloji, Ankara
  - Ankara Sehir Hastanesi Cardiology, Ankara
  - Bursa Şehir Hastanesi- Kardiyoloji, Bursa
  - Trakya University, Edirne
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul
  - Erciyes University Cardiology, Kayseri
  - Erciyes Üniversitesi Hastanesi- Kardiyoloji, Kayseri
  - Kocaeli Üniversitesi Hastanesi- Kardiyoloji, Kocaeli
- United Kingdom (5):
  - Raigmore Hospital, Inverness, Highland
  - St. Richard's Hospital_Cardiology, Chichester, West Sussex
  - FutureMeds, Birmingham
  - Ninewells Hospital, Dundee
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com